CLINICAL TRIAL: NCT05963997
Title: A Phase 1b/2 Open-label Study of Samuraciclib in Combination With Elacestrant in Participants With Metastatic or Locally Advanced Hormone Receptor-positive and Human Epidermal Growth Factor Receptor 2-negative Breast Cancer
Brief Title: A Study of Samuraciclib and Elacestrant in Participants With Metastatic or Locally Advanced HR+/HER2-negative Breast Cancer
Acronym: SUMIT-ELA
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Carrick Therapeutics Limited (Industry)
Collaborators: Berlin-Chemie AG Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CT7001_003; 2023-503846-30-00 (Registry Identifier: EU CTIS); 2023-000072-35 (EudraCT Number)
Record Dates: First submitted 2023-06-30; First posted 2023-07-27 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Breast Cancer; Locally Advanced Breast Cancer; Breast Cancer
Keywords: Metastatic Breast Cancer; Advanced Breast Cancer; Breast Cancer; HR Positive; HER2-Negative
MeSH Terms: conditions — Breast Neoplasms | interventions — RAD1901

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Up to 6 evaluable participants will receive samuraciclib 240 mg in combination with elacestrant 300 mg in cycles of 28 days (Cycle 1 to 6), 56 days (Cycle 7 to 9) and up to 84 days (Cycles 10 onwards).
  Interventions: Drug: Samuraciclib; Drug: Elacestrant Dihydrochloride
- Cohort 2 (Experimental): Up to 6 evaluable participants will receive samuraciclib in combination with elacestrant at the SRC recommended dose (anticipated 360mg samuraciclib, 300 mg elacestrant) in cycles of 28 days (Cycle 1 to 6), 56 days (Cycle 7 to 9) and up to 84 days (Cycles 10 onward).
  Interventions: Drug: Samuraciclib; Drug: Elacestrant Dihydrochloride
- Cohort 3 (Experimental): Up to 6 evaluable participants will receive samuraciclib in combination with elacestrant at the SRC recommended dose (anticipated 360mg samuraciclib, 400 mg elacestrant) in cycles of 28 days (Cycle 1 to 6), 56 days (Cycle 7 to 9) and up to 84 days (Cycles 10 onward).
  Interventions: Drug: Samuraciclib; Drug: Elacestrant Dihydrochloride
- Cohort 4 Expansion (Experimental): Up to 30 evaluable participants will receive samuraciclib in combination with elacestrant at the SRC recommended dose (anticipated 360mg samuraciclib, 400 mg elacestrant) in cycles of 28 days (Cycle 1 to 6), 56 days (Cycle 7 to 9) and up to 84 days (Cycles 10 onward).
  Interventions: Drug: Samuraciclib; Drug: Elacestrant Dihydrochloride

INTERVENTIONS:
Drug: Samuraciclib — Samuraciclib capsules by mouth once a day
Drug: Elacestrant Dihydrochloride — Elacestrant tablets by mouth once a day
  Other Names: ORSERDU

SUMMARY:
This is an international, multisite, open-label, Phase 1b/2 study, to confirm safety and efficacy of samuraciclib in combination with elacestrant in adult participants with metastatic or locally advanced Hormone Receptor (HR) positive and Human Epidermal Growth Factor Receptor (HER)2-negative breast cancer.

DETAILED DESCRIPTION:
This is a multiple cohort study, an initial dose escalation phase is designed to confirm the safe dose of samuraciclib in combination with elacestrant. A Safety Review Committee (SRC) will monitor the safety, tolerability, and PK data during this phase. Once ascertained, an expansion cohort will be opened to explore the efficacy of samuraciclib in combination with elacestrant.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of ER-positive, HER2-negative locally advanced or metastatic breast cancer.
* Documented objective disease progression while on or within 6 months after the end of the most recent therapy.
* Received prior AI in combination with a CDK4/6i as the last therapy
* Known TP53 and ESR1 mutation status.
* Participants must have measurable disease or bone only disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
* Pre/peri-menopausal participants must have commenced treatment with a luteinizing hormone-releasing hormone (LHRH) agonist at least 4 weeks prior to first dose of study intervention.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1 with no deterioration over the past 2 weeks.
* Expected life expectancy of >12 weeks in the judgement of the treating investigator.

Exclusion Criteria:

* Inflammatory breast cancer.
* Participants with any other active malignancy within 3 years prior to enrollment, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix.
* More than 1 line of endocrine treatment for locally advanced or metastatic disease treatment.
* Inadequate hepatic, renal, and bone marrow function.
* Clinically significant cardiovascular disease.
* Any current or prior central nervous system metastases, carcinomatous meningitis, or leptomeningeal disease.
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Phase 1b (Dose-finding) | From the date of first dose of any study intervention (Day 1 Cycle 1) and through 28 days after the last dose of any study intervention
  Identification of Samuraciclib + Elacestrant combination, Phase 2, expansion dose level.
  Incidence and severity of adverse events as graded by the National Cancer Institute Common Terminology Criteria for Adverse events (NCI-CTCAE) v5.0. Safety will be assessed by monitoring treatment - emerged severe and dose limiting adverse events and clinically relevant changes in vital signs and clinical laboratory results
Phase 2 (Expansion) | From the date of first dose of any study intervention (Cycle 1 Day 1) until the first documentation of disease progression, death, withdrawal of consent, or start of new anticancer therapy (assessed up to week 48)
  Progression Free Survival (PFS) is defined as the time from the date of first dose of IMP (Cycle 1 Day 1) to the date of the first documentation of objective progressive disease (PD) or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Treatment-Emergent Adverse Events and Laboratory Abnormalities (Safety and Tolerability) | From the date of first dose of any study intervention through 28 days after the last dose of any study intervention
  Type, incidence, severity (as graded by CTCAE v5.0), seriousness and relationship to study medications of AEs and any laboratory abnormalities. Safety will be assessed by monitoring adverse events and clinically relevant changes in vital signs and clinical laboratory results.
Clinical Benefit Response (CBR) | From the date of first dose of any study intervention (Cycle 1 Day 1) to ≥ 24 weeks or until disease progression or death to any cause (assessed up to week 24)
  CBR is defined as the overall complete response (CR), partial response (PR), or stable disease (SD) ≥ 24 weeks according to RECIST version 1.1 recorded from enrolment until disease progression, or death due to any cause.
Overall response rate (ORR) | the date of first dose of study intervention (Cycle 1 Day 1) until the first documentation of disease progression, death, withdrawal of consent, or start of new anticancer therapy (assessed up to week 48)
  ORR is defined as the proportion of participants with a reduction in tumor burden with CR or PR according to RECIST version 1.1.
  ORR will be estimated for participants who received at least 1 dose of IMP, had measurable disease at baseline and had a postbaseline tumor assessment.
Duration of Response (DOR) | From the date of first dose of study intervention (Cycle 1 Day 1) until the first documentation of disease progression, death, withdrawal of consent, or start of new anticancer therapy (assessed up to week 48)
  DOR is defined as the time from the date of first documentation of objective tumor response (CR or PR) to the earliest documented disease progression per RECIST version 1.1
Best percent change in tumor size. | From the date of first dose of study intervention (Cycle 1 Day 1) until the first documentation of disease progression, death, withdrawal of consent, or start of new anticancer therapy (assessed up to week 48)
  Best percent change in tumor size is defined as the percentage change in the sum of the longest diameters of target lesions
Samuraciclib plasma exposure: Cmax | Day 1 of Cycles 1 and Cycle 2 (each cycle is 28 days)
  Plasma concentration for Samuraciclib
Elacestrant exposure: Cmax | Day 1 of Cycles 1 and Cycle 2 (each cycle is 28 days)
  Plasma concentrations for Elacestrant
Samuraciclib plasma exposure: Ctrough | Cycle 1 Day 2 and 15; Day 2 of Cycle 2; Day 1 of Cycles 3-6 and end of treatment within 28 days of last dose of IMP and prior to the initiation of a new anticancer therapy (each cycle is 28 days)]
Elacestrant exposure: Ctrough | Cycle 1 Day 2 and Day 15; Cycle 2 Day 2 of Cycle 2 and Day 1 of Cycles 3-6 and at end of treatment within 28 days of the last dose of IMP and prior to the initiation of a new anticancer therapy (each cycle is 28 days)
Genotyping for ESR1 and TP53 mutations | Screening
  Genotyping for ESR1 and TP53 mutations to evaluate correlations between ESR1 and TP53 mutations and efficacy/safety findings

CONTACTS AND LOCATIONS:
Locations (23):
- United States (5):
  - Site 38 - Northwestern University, Feinberg School of Medicine, Northwestern University, Chicago, Illinois
  - Site 42 - Dana-Farber Cancer Institute, EDDC, Boston, Massachusetts
  - Site 35 - Cleveland Clinic, Taussig Cancer Institute, Cleveland, Ohio
  - Site 41 - The START Center for Cancer Care, South Texas Oncology and Hematology, San Antonio, Texas
  - Site 32 - Swedish Medical Center, Swedish Cancer Institute (SCI),Cherry Hill Campus, Seattle, Washington
- France (5):
  - Site 81 - Bergonie unicancer, Nouvelle-Aquitaine, L'Institut Bergonie, Bordeaux
  - Site 80 - Centre Jean Bernard, Clinique Victor Hugo, Le Mans
  - Site 83 - Institut Paoli Calmettes (IPC), Marseille
  - Site 85 - Institut Curie, Paris
  - Site 82 - Institut de Cancerologie de Ouest (ICO), Saint-Herblain
- Spain (10):
  - Site 65 - Complexo Hospitalario Universitario A Coruña, A Coruña
  - Site 64 - Hospital Clinic de Barcelona (Hospital Clinic i Provincial), Barcelona
  - Site 68 -Hospital Universitario Vall d'Hebron, Barcelona
  - Site 61 - Institut Catala d'Oncologia (ICO), Hospital Duran i Reynals Location, L'Hospitalet de Llobregat
  - Site 62 - Universidad de Navarra, Clinica Universidad de Navarra (CUN), Madrid
  - Site 63 - South Texas Accelerated Research Therapeutics, CIOCC, Hospital Madrid Norte-Sanchinarro, Madrid
  - Site 66 - Hospital Clinico San Carlos, Madrid
  - Site 69 - Universidad de Navarra - Clinica Universidad de Navarra (CUN), Pamplona
  - Site 60 - NEXT Oncology EU Hospital Universitario Quiron Salud Madrid, Pozuelo de Alarcón
  - Site 67 - Universidad de Sevilla, Hospital Universitario Virgen Macarena, Seville
- United Kingdom (3):
  - Site 12 - Belfast City Hospital, Belfast
  - Site 4 - The Christie NHS Foundation Trust, Manchester
  - Site 2 - Oxford University Hospitals NHS Trust - Churchill Hospital, Oxford